CLINICAL TRIAL: NCT00554645
Title: Multi-Disciplinary Group Intervention Versus Traditional Information Towards Severely Overweight Children and Their Families -
Brief Title: GRIB Forsoeget-2004
Acronym: GRIB-2004
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Forskningspuljen (Other Government)
Collaborators: Den Sundhedsvidenskabelige Forskningsfond (Region 3) (Unknown); Østdansk Sundhedsvidenskabeligt Forskningsforums Konsuletttjeneste (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ø-2003-1-40
Record Dates: First submitted 2007-11-05; First posted 2007-11-07 (Estimated); Last update posted 2007-11-07 (Estimated); Status verified 2007-11

CONDITIONS: Overweight
Keywords: obesity; children; psychological intervention
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Multi-disciplinary group intervention
  Interventions: Behavioral: multi-disciplinary group intervention
- 2 (Active Comparator): traditional information
  Interventions: Other: traditional information

INTERVENTIONS:
Behavioral: multi-disciplinary group intervention — children:weekley session in 6 months, monthly sessions for 6 months parents: bi-monthly sessions for 6 months, monthly sessions for 6 months
  Arms: 1
Other: traditional information — 1 session of nutritional advise for parents and child and 1 follow-up after one month
  Arms: 2

SUMMARY:
The difficulties in loosing weight may not stem from lack og knowledge about nutrition, as implied by the standard treatment but from difficulties in following the advice. The hypothesis is, that revealing and addressing these difficulties psychotherapeutically may be more efficient in obtaining weight reduction. The effect of psychological group treatment of severely overweight children and their parents is compared with traditional nutritional information. In other words: Which is better: back-up or enlightenment?

DETAILED DESCRIPTION:
At on-set the children get a medical examination, blood-tests, measurement of height, weight, skin-fold, waist and hip. Children and parents fill out questionnaires on social and educational background as well as motivation and expectations to the treatment. All Children are thereafter randomised into two groups:multi-disciplinary group intervention versus traditional information. The randomisation is stratified according to gender and degree of overweight (135%-145% and >145%) supposing that the degree of overweight may mirror the difficulties in loosing weight. The experimental intervention consists of one lecture of general nutrition, weekly psychological group sessions for the children followed by physical exercise, and separate bi-monthly group sessions for the parents. After six months children and parents go to separate group sessions once a month for six months. The control group is offered nutritional advice once with a brief follow-up after one month. The height and weight of the children is measured every month, and the fat % is measured with DEXA-scanning at on-set, after six months, and after twelve months

ELIGIBILITY:
Inclusion Criteria:

* Weight compared to hight over 135% of the Danish norms (www.peadiatri.dk)

Exclusion Criteria:

* None of the parents wants to participate
* Diagnosed somatic course of overweight
* Parents or children do not speak danish
* Sever physical handicap
* Psychiatric illness or mental retardation in children or parents
* Severe child abuse
* Siblings participation in the trail.

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2004-01; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Body Mass Index | Baseline, 6 months, 12 months

SECONDARY OUTCOMES:
fat% measured by DEXA scan, Hip/waist ratio, skinfold | Baseline, 6 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ole Andersen, dr. med., Study Chair — former chief administration physician, peadiatrisk Enhed, Hilleroed Sygehus, 3400 Hilleroed
Locations (1):
- Peaditrisk enhed, Helse vej 2, Hilleroed, Regionh, Denmark